CLINICAL TRIAL: NCT00394173
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group, Multicenter Study to Evaluate the Efficacy and Safety of DNK333 25mg b.i.d. Given Orally for 4 Weeks in Female Patients With Diarrhea-predominant Irritable Bowel Syndrome (IBS-D)
Brief Title: Efficacy, Safety and Tolerability of DNK333 (25 mg Bid) in Women With Diarrhea-predominant Irritable Bowel Syndrome (IBS-D)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CDNK333B2202
Record Dates: First submitted 2006-10-30; First posted 2006-10-31 (Estimated); Last update posted 2017-02-27 (Actual); Status verified 2017-02

CONDITIONS: Irritable Bowel Syndrome With Diarrhea (IBS-D)
Keywords: IBS; diarrhea; gastrointestinal functional disorder; IBS-D
MeSH Terms: conditions — Diarrhea; Gastrointestinal Diseases | interventions — DNK 333

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: DNK333
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DNK333 — DNK333 25mg b.i.d. given orally for 4 weeks
  Arms: 1
Drug: Placebo — Matching placebo
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the efficacy of DNK333 compared to placebo for relieving symptoms of IBS-D in female patients.

ELIGIBILITY:
Inclusion criteria:

* Women of 18 - 65 years of age with IBS-D as defined by the Rome II criteria.
* The Rome II criteria is a system used for diagnosing functional gastrointestinal disorders such as irritable bowel syndrome. It involves completing of a questionnaire about gastrointestinal symptoms.
* Patients who are 50 years of age and older must have had a colonoscopy OR a flexible sigmoidoscopy plus a double-contrast barium enema within the past 5 years, which demonstrated no clinically significant findings.
* Clinically significant findings may include but are not limited to malignant tumors, multiple (≥3) or advanced adenomas, inflammatory bowel disease, diverticulitis, ischaemic colitis, lymphocytic colitis, or collagenous colitis.
* Patients must report ≥ 3 days with IBS-related abdominal pain/discomfort plus at least 3 days of 2 or more of the following events during the baseline period:
* ≥ 3 bowel movements/day
* Bowel urgency
* Loose or watery stool

Exclusion Criteria:

* Patients who answer "yes" to either or both of the two weekly satisfaction questions during the baseline period. The questions are: (1) Over the past week did you have satisfactory relief of your IBS-related abdominal pain/discomfort? (2) Over the last week did you have satisfactory relief of your overall IBS-D symptoms?
* Patients with hard or lumpy stools for more than one day during the baseline period.
* Lactose intolerant patients relieved on a lactose free diet.
* Use of antidepressants (tricyclic, SSRI etc), opioid analgesic drugs or drugs specifically affecting bowel motility during the course of the trial.
* Women of child-bearing potential who do not use an acceptable methods of contraception.
* Pregnant or nursing (lactating) women.

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: Female
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2006-09; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Satisfactory relief of IBS-related abdominal pain/discomfort | 4 weeks
Satisfactory relief of overall IBS-D symptoms | 4 weeks

SECONDARY OUTCOMES:
Occurrence and control of bowel urgency | 4 weeks
Change in stool frequency | 4 weeks
Severity of abdominal bloating | 4 weeks
Severity of abdominal pain/discomfort | 4 weeks
Safety | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals Corp., Study Chair — NPC
Locations (43):
- United States (37):
  - Investigative Site, Tucson, Arizona
  - Investigative Site, North Little Rock, Arkansas
  - Investigative Site, Los Angeles, California
  - Investigative Site, Orange, California
  - Investigative Site, Riverside, California
  - Investigative Site, Sacramento, California
  - Investigative Site, San Diego, California
  - Investigative Site, Colorado Springs, Colorado
  - Investigative Site, Bristol, Connecticut
  - Investigative Site, Hartford, Connecticut
  - Investigative Site, Boca Raton, Florida
  - Investigative Site, Gainesville, Florida
  - Investigative Site, Hollywood, Florida
  - Investigative Site, Jacksonville, Florida
  - Investigative Site, Miami, Florida
  - Investigative Site, New Smyrna Beach, Florida
  - Investigative Site, Tampa, Florida
  - Investigative Site, Arlington Heights, Illinois
  - Investigative Site, Rockford, Illinois
  - Investigative Site, Boston, Massachusetts
  - Investigative Site, Wellesley Hills, Massachusetts
  - Investigative Site, Mexico, Missouri
  - Investigative Site, Buffalo, New York
  - Investigative Site, Great Neck, New York
  - Investigative Site, Elkin, North Carolina
  - Investigative Site, Cincinnati, Ohio
  - Investigative Site, Oklahoma City, Oklahoma
  - Investigative Site, Portland, Oregon
  - Investigative Site, Chattanooga, Tennessee
  - Investigative Site, Lake Jackson, Texas
  - Investigative Site, San Antonio, Texas
  - Investigative Site, Salt Lake City, Utah
  - Investigative Site, Chesapeake, Virginia
  - Investigative Site, Bellevue, Washington
  - Investigative Site, Everett, Washington
  - Investigative Site, Monroe, Washington
  - Investigative Site, Seattle, Washington
- Canada (6):
  - Investigative Site, Calgary, Alberta
  - Investigative Site, St. John's, Newfoundland and Labrador
  - Investigative Site, Hamilton, Ontario
  - Investigative Site, Montreal, Quebec
  - Investigative Site, Québec, Quebec
  - Investigative Site, Sherbrooke, Quebec

REFERENCES:
- [Result] Zakko S, Barton G, Weber E, Dunger-Baldauf C, Ruhl A. Randomised clinical trial: the clinical effects of a novel neurokinin receptor antagonist, DNK333, in women with diarrhoea-predominant irritable bowel syndrome. Aliment Pharmacol Ther. 2011 Jun;33(12):1311-21. doi: 10.1111/j.1365-2036.2011.04656.x. Epub 2011 Apr 20. PMID 21507028